CLINICAL TRIAL: NCT03755934
Title: A Randomised, Double-Blind, Placebo-Controlled, Dose-Response Study of the Efficacy and Safety of MEDI7352 in Subjects With Painful Diabetic Neuropathy
Brief Title: Efficacy and Safety of MEDI7352 in Participants With Painful Diabetic Neuropathy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was prematurely terminated due to longer enrolment time than was anticipated.
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D5680C00002; 2018-002523-42 (EudraCT Number)
Record Dates: First submitted 2018-10-31; First posted 2018-11-28 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Painful Diabetic Neuropathy
MeSH Terms: conditions — Diabetic Neuropathies

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double blind
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Placebo (Placebo Comparator): Participants received 6 doses of intravenous (IV) placebo infusion matched to MEDl7352 during 12-week treatment period.
  Interventions: Other: Placebo
- MEDl7352 Low Dose (Experimental): Participants received 6 doses of IV MEDl7352 low dose during 12-week treatment period.
  Interventions: Drug: MEDI7352
- MEDl7352 Medium Dose (Experimental): Participants received 6 doses of IV MEDl7352 medium dose during 12-week treatment period.
  Interventions: Drug: MEDI7352
- MEDI7352 High Dose (Experimental): Participants received 6 doses of IV MEDl7352 high dose during 12-week treatment period.
  Interventions: Drug: MEDI7352

INTERVENTIONS:
Drug: MEDI7352 — Participants will receive IV infusion of MEDI7352 as stated in arm description.
  Arms: MEDI7352 High Dose; MEDl7352 Low Dose; MEDl7352 Medium Dose
Other: Placebo — Participants will receive IV infusion of placebo as stated in arm description.
  Arms: Placebo

SUMMARY:
This is a study investigating the effect of MEDI7352 on chronic pain in participants with painful diabetic neuropathy.

The study incudes a screening period of up to 45 days and a 12-week treatment period during which MEDI7352 or placebo will be administered intravenously (IV) on 6 occasions, with each dose separated by 14 days. There will be a 6-week follow-up period.

Participants will randomly be assigned to double-blind treatment with one of 4 dose levels of MEDI7352 or placebo.

ELIGIBILITY:
Key Inclusion criteria:

* Male, or postmenopausal or surgically sterile female, 18 to 80 years of age
* Body mass index of ≤ 42 kg/m^2.
* Chronic painful diabetic neuropathy (PDN) persistent for 6 months or longer, not adequately controlled by standard of care treatments.
* Mean pain intensity score of ≥ 4, as measured on an 11-point (0-10) numerical rating scale (NRS).
* Willing and able to discontinue all non-steroidal anti-inflammatory drug (NSAID) or cyclooxygenase-2 (COX-2) analgesic therapy.
* Currently be taking medication for the treatment of PDN. Participants should be taking at least one of the first-line medications (consistent with regional or local standard of care guidelines for PDN).

Key Exclusion criteria:

* Presence of other clinically significant neuropathy (eg, hereditary neuropathy, inflammatory neuropathy) or other clinically significant disorder (eg, nerve compression injury) involving abnormal peripheral sensation, with an aetiology that is considered to be distinct from that of PDN, and that is likely to interfere with assessment of peripheral nerve function, as judged by the investigator.
* History of osteonecrosis, rapidly progressing osteoarthritis (OA), subchondral insufficiency fractures, neurogenic arthropathy, or analgesia-induced arthropathy.
* Diagnosis of clinically significant OA currently affecting a major joint in the upper extremity (shoulder, elbow, or wrist) or lower extremity (hip, knee, or ankle) or axial spine; or other degenerative disease affecting any joint in participants for whom, in the opinion of the investigator, there is an identified risk of osteonecrosis, rapidly progressing OA, subchondral insufficiency fractures, neurogenic arthropathy, or analgesia-induced arthropathy.
* Chronic pain condition, other than PDN, that is likely to interfere with the evaluation of the participant's PDN pain, as judged by the investigator.
* Haemoglobin A1C greater than 10.0% (> 10.0%).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2018-11-19 (Actual); Primary Completion 2023-06-29 (Actual); Study Completion 2023-06-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (28):
- Research Site, Gentofte Municipality, Denmark
- Hungary (2):
  - Research Site, Balatonfüred
  - Research Site, Budapest
- Poland (11):
  - Research Site, Bydgoszcz
  - Research Site, Gdansk
  - Research Site, Katowice
  - Research Site, Krakow
  - Research Site, Lublin
  - Research Site, Olsztyn
  - Research Site, Poznan
  - Research Site, Sochaczew
  - Research Site, Torun
  - Research Site, Warsaw
  - Research Site, Wroclaw
- Romania (5):
  - Research Site, Bucharest
  - Research Site, Călăraşi
  - Research Site, Craiova
  - Research Site, Galati
  - Research Site, Târgu Mureş
- United Kingdom (9):
  - Research Site, Barnsley
  - Research Site, Blackpool
  - Research Site, Cannock
  - Research Site, Cardiff
  - Research Site, Leeds
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Prescot
  - Research Site, Stockton-on-Tees

REFERENCES:
- See also: CSR synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5680C00002&attachmentIdentifier=047c595c-3112-4e4f-972f-f0ff1c0af44f&fileName=synopsis-Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 45 sites in 4 countries (the United Kingdom, Hungary, Poland, and Romania).
Pre-assignment Details: A total of 112 participants were randomized, of which 107 participants received at least one dose of study drug.
Groups:
- MEDl7352 Low Dose; MEDl7352 Meduim Dose; MEDI7352 High Dose: Participants received 6 doses of IV MEDl7352 during 12-week treatment period.
Period: Overall Study
Arm/Group | Placebo | MEDl7352 Low Dose | MEDl7352 Meduim Dose | MEDI7352 High Dose
Started | 54 | 6 | 16 | 36
Treated | 54 | 4 | 14 | 35
Completed | 40 | 4 | 12 | 30
Not Completed | 14 | 2 | 4 | 6
Not completed — Adverse Event | 4 | 1 | 1 | 3
Not completed — Physician Decision | 2 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 5 | 0 | 0 | 1
Not completed — Other | 3 | 1 | 3 | 1

BASELINE CHARACTERISTICS:
Population: The Screening Population includes all participants who were enrolled and provided informed consent and demographic and/or baseline screening assessments.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | MEDl7352 Low Dose | MEDl7352 Meduim Dose | MEDI7352 High Dose | Total
Number analyzed (Participants) | 54 | 6 | 16 | 36 | 112
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.7 (8.02) | 60.7 (17.14) | 60.1 (11.49) | 60.1 (10.21) | 60.4 (9.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 0 | 5 | 15 | 40
  Male | 34 | 6 | 11 | 21 | 72
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 54 | 6 | 16 | 36 | 112
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 2 | 0 | 2
  White | 53 | 6 | 14 | 36 | 109
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Weekly Average of Average Daily Pain Score to Week 12
Description: Change from baseline to Week 12 in weekly average of average daily pain score is reported. Participants assessed their perceived daily average neuropathic pain over the previous 24 hours using an 11-point numerical rating scale (NRS), with 0 representing no pain and 10 representing the worst pain imaginable. Participants were instructed to assess their average daily pain at approximately the same time every morning, and to record the response in a subject diary (electronic patient-reported outcome [ePRO]).
Time Frame: Baseline (Day -7 to Day -1, inclusive) through Week 12
Population: Modified intent-to-treat (mITT) population included all participants who received at least 1 dose of any double-blind study drug and have at least 1 daily NRS assessment while receiving the treatment.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | MEDl7352 Low Dose | MEDl7352 Meduim Dose | MEDI7352 High Dose
Number analyzed (Participants) | 54 | 4 | 14 | 35
Units on a scale | -1.244 (1.7327) | -3.387 (1.9605) | -0.615 (1.0431) | -2.699 (2.0819)
Statistical Analysis 1: Comparison: Placebo vs MEDl7352 Low Dose; Test type: Superiority; p = 0.0437, ANCOVA — ANCOVA by dose using NRS baseline value and co-medication as covariates, with CFB to Week 12 (LOCF) as dependent variable was used to derive p-value; LS mean estimate = -1.96, 95% CI 2-sided [-3.87 to -0.06], Standard Error of Mean 0.961
Statistical Analysis 2: Comparison: Placebo vs MEDl7352 Meduim Dose; Test type: Superiority; p = 0.1878, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LS mean estimate = 0.72, 95% CI 2-sided [-0.36 to 1.79], Standard Error of Mean 0.541
Statistical Analysis 3: Comparison: Placebo vs MEDI7352 High Dose; Test type: Superiority; p = 0.0009, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LS mean estimate = -1.39, 95% CI 2-sided [-2.19 to -0.58], Standard Error of Mean 0.407

2. Secondary Outcome: Change From Baseline in Weekly Average of Average Daily Pain Score
Description: Change from baseline to Weeks 2, 4, 6, 8, 10, and 18 in weekly average of average daily pain score is reported. Participants assessed their perceived daily average neuropathic pain over the previous 24 hours using an 11-point NRS, with 0 representing no pain and 10 representing the worst pain imaginable. Participants were instructed to assess their average daily pain at approximately the same time every morning, and to record the response in a subject diary (ePRO).
Time Frame: Baseline (Day -7 to Day -1, inclusive), Weeks 2, 4, 6, 8, 10, and 18
Population: mITT population included all participants who received at least 1 dose of any double-blind study drug and have at least 1 daily NRS assessment while receiving the treatment. Here, number analyzed (n) denotes those participants who were evaluable at the specified time point.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | MEDl7352 Low Dose | MEDl7352 Meduim Dose | MEDI7352 High Dose
Number analyzed (Participants) | 54 | 4 | 14 | 35
Units on a scale
  Week 2: number analyzed (Participants) | 53 | 4 | 14 | 35
  Week 2 | -0.385 (0.6863) | -1.089 (1.0258) | -0.311 (0.6285) | -0.540 (1.2503)
  Week 4: number analyzed (Participants) | 54 | 4 | 13 | 35
  Week 4 | -0.563 (1.0173) | -2.173 (1.4266) | -0.144 (0.9143) | -1.508 (1.5130)
  Week 6: number analyzed (Participants) | 50 | 4 | 13 | 34
  Week 6 | -0.955 (1.3236) | -2.458 (2.2156) | -0.578 (1.0715) | -2.044 (1.7916)
  Week 8: number analyzed (Participants) | 46 | 4 | 12 | 33
  Week 8 | -1.236 (1.6026) | -2.393 (2.0249) | -0.690 (1.2819) | -2.372 (2.0607)
  Week 10: number analyzed (Participants) | 44 | 4 | 12 | 33
  Week 10 | -1.418 (1.6274) | -2.595 (2.2003) | -0.712 (1.2164) | -2.629 (1.9943)
  Week 18: number analyzed (Participants) | 40 | 4 | 12 | 30
  Week 18 | -1.764 (1.8415) | -2.607 (2.2020) | -0.550 (1.2333) | -2.559 (2.1241)

3. Secondary Outcome: Percentage of Participants With >= 30% and >= 50% Reductions in Weekly Average of Average Daily Pain Score
Description: Percentage of participants with >= 30% and >= 50% decrease in weekly average of average daily pain score from baseline is reported. Participants assessed their perceived daily average neuropathic pain over the previous 24 hours using an 11-point NRS, with 0 representing no pain and 10 representing the worst pain imaginable. Participants were instructed to assess their average daily pain at approximately the same time every morning, and to record the response in a subject diary (ePRO).
Time Frame: Baseline (Day -7 to Day -1, inclusive), Weeks 4, 8, 12, and 18 (follow-up)
Population: mITT population included all participants who received at least 1 dose of any double-blind study drug and have at least 1 daily NRS assessment while receiving the treatment. Here, number of participants analyzed (N) denotes those participants who were evaluable for the specified outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | MEDl7352 Low Dose | MEDl7352 Meduim Dose | MEDI7352 High Dose
Number analyzed (Participants) | 54 | 4 | 13 | 35
Percentage of participants
  >=30%: Week 4 | 3.7 | 75.0 | 7.7 | 34.3
  >=30%: Week 8: number analyzed (Participants) | 46 | 4 | 12 | 33
  >=30%: Week 8 | 28.3 | 75.0 | 16.7 | 57.6
  >=30%: Week 12: number analyzed (Participants) | 43 | 4 | 12 | 33
  >=30%: Week 12 | 32.6 | 75.0 | 8.3 | 66.7
  >=30%: Week 18: number analyzed (Participants) | 40 | 4 | 12 | 30
  >=30%: Week 18 | 35.0 | 50.0 | 25.0 | 56.7
  >=50%: Week 4 | 1.9 | 0 | 0 | 14.3
  >=50%: Week 8: number analyzed (Participants) | 46 | 4 | 12 | 33
  >=50%: Week 8 | 13.0 | 25.0 | 8.3 | 36.4
  >=50%: Week 12: number analyzed (Participants) | 43 | 4 | 12 | 33
  >=50%: Week 12 | 11.6 | 50.0 | 8.3 | 42.4
  >=50%: Week 18: number analyzed (Participants) | 40 | 4 | 12 | 30
  >=50%: Week 18 | 15.0 | 25.0 | 0 | 40.0

4. Secondary Outcome: Change From Baseline in Galer Neuropathic Pain Scale (NPS)
Description: Participants were assessed for their neuropathic pain using the Galer NPS, which included 2 descriptors of pain, including intensity and unpleasantness, and 8 descriptors that assessed specific qualities of neuropathic pain: sharp, hot, dull, cold, sensitive, itchy, deep, and surface pain. Each of these 10 dimensions had a 0 to 10 NRS in which 0 is equal to no pain and 10 equals most intense pain. Galer NPS total score (ranges from 0 to 100; with 0 and 100 representing the no and highest degree of neuropathic-like symptoms, respectively) is sum of pain intensity, pain unpleasantness, pain sharpness, pain hotness, pain dullness, pain coldness, pain sensitivity, pain itching, deep pain intensity, and surface pain intensity (all in an 11-point NRS). Change from baseline to Weeks 4, 8, 12, and 18 (follow-up) in Galer NPS total score is reported.
Time Frame: Baseline (Day -7 to Day -1, inclusive), Weeks 4, 8, 12, and 18 (follow-up)
Population: mITT population included all participants who received at least 1 dose of any double-blind study drug and have at least 1 daily NRS assessment while receiving the treatment. Number of participants analyzed (N) denotes the number of participants evaluated for this outcome measure. Here, number analyzed (n) denotes those participants who were evaluable at the specified time point.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | MEDl7352 Low Dose | MEDl7352 Meduim Dose | MEDI7352 High Dose
Number analyzed (Participants) | 48 | 4 | 12 | 31
Units on a scale
  Week 4: number analyzed (Participants) | 48 | 4 | 11 | 31
  Week 4 | -13.333 (29.0461) | -5.750 (10.5317) | -10.727 (21.3967) | -26.387 (26.9922)
  Week 8: number analyzed (Participants) | 44 | 4 | 12 | 31
  Week 8 | -19.136 (31.5577) | -8.750 (18.2094) | -19.333 (23.7538) | -29.516 (32.3140)
  Week 12: number analyzed (Participants) | 39 | 4 | 11 | 29
  Week 12 | -24.385 (31.1081) | -28.750 (16.6808) | -22.000 (28.9379) | -34.586 (31.2622)
  Week 18 (follow-up): number analyzed (Participants) | 36 | 4 | 11 | 29
  Week 18 (follow-up) | -25.722 (33.6151) | -23.000 (23.3095) | -27.909 (30.3725) | -25.414 (25.8947)

5. Secondary Outcome: Change From Baseline in Daily Sleep Interference Scale (DSIS)
Description: Participants were assessed for how their neuropathic pain interferes with their sleep using the DSIS. It has an 11 point Likert response scale (0-10) that asked participants to "select the number that best describes how much your pain has interfered with your sleep during the past 24 hours". Responses vary from 0 (did not interfere with sleep) to 10 (completely interfered with sleep-unable to sleep due to pain). The DSIS was completed by participants once a day (upon awakening) to accurately capture variability in sleep interference due to pain on a daily basis, thus minimizing recall bias. Change from baseline to Weeks 4, 8, 12, and 18 (follow-up) in DSIS is reported.
Time Frame: Baseline (Day -7 to Day -1, inclusive), Weeks 4, 8, 12, and 18 (follow-up)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | MEDl7352 Low Dose | MEDl7352 Meduim Dose | MEDI7352 High Dose
Number analyzed (Participants) | 52 | 4 | 13 | 35
Units on a scale
  Week 4 | -0.760 (1.1212) | -2.810 (2.6979) | -0.979 (1.7930) | -1.790 (1.5688)
  Week 8: number analyzed (Participants) | 46 | 4 | 12 | 33
  Week 8 | -1.417 (1.7654) | -3.143 (2.7430) | -1.127 (1.4907) | -2.373 (2.1368)
  Week 12: number analyzed (Participants) | 42 | 4 | 12 | 33
  Week 12 | -1.668 (2.1928) | -3.735 (2.7598) | -1.077 (1.4769) | -2.725 (2.2484)
  Week 18 (follow-up): number analyzed (Participants) | 40 | 4 | 12 | 30
  Week 18 (follow-up) | -1.824 (2.2582) | -3.036 (2.6557) | -0.865 (1.2795) | -2.602 (2.4427)

6. Secondary Outcome: Percentage of Participants With 'Improved', 'Much Improved', or 'Very Much Improved' Status in Patient Global Impression of Change (PGIC)
Description: Participants rated their overall improvement in health status using the PGIC. The PGIC consisted of a 7-point scale where 1 = very much improved and 7 = very much worse. The participants were asked the following question: How would you rate your overall improvement with treatment during the clinical study?, where the response options included the following: Very Much Improved, Much Improved, Minimally Improved, No Change, Minimally Worse, Much Worse, and Very Much Worse.
Time Frame: Baseline (Day -7 to Day -1, inclusive), Weeks 4, 8, 12, and 18 (follow-up)
Population: mITT population included all participants who received at least 1 dose of any double-blind study drug and have at least 1 daily NRS assessment while receiving the treatment. Number of participants analyzed (N) denotes the number of participants who were PGIC responders. Here, number analyzed (n) denotes those participants who were evaluable at the specified time point.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | MEDl7352 Low Dose | MEDl7352 Meduim Dose | MEDI7352 High Dose
Number analyzed (Participants) | 48 | 4 | 12 | 31
Percentage of participants
  Week 4: Improved: number analyzed (Participants) | 48 | 4 | 11 | 31
  Week 4: Improved | 50.0 | 50.0 | 45.5 | 41.9
  Week 4: Much Improved: number analyzed (Participants) | 48 | 4 | 11 | 31
  Week 4: Much Improved | 2.1 | 25.0 | 27.3 | 29.0
  Week 4: Very Much Improved: number analyzed (Participants) | 48 | 4 | 11 | 31
  Week 4: Very Much Improved | 2.1 | 0 | 0 | 6.5
  Week 8: Improved: number analyzed (Participants) | 44 | 4 | 12 | 31
  Week 8: Improved | 36.4 | 25.0 | 58.3 | 41.9
  Week 8: Much Improved: number analyzed (Participants) | 44 | 4 | 12 | 31
  Week 8: Much Improved | 31.8 | 50.0 | 41.7 | 38.7
  Week 8: Very Much Improved: number analyzed (Participants) | 44 | 4 | 12 | 31
  Week 8: Very Much Improved | 2.3 | 0 | 0 | 6.5
  Week 12: Improved: number analyzed (Participants) | 39 | 4 | 11 | 29
  Week 12: Improved | 48.7 | 0 | 54.5 | 44.8
  Week 12: Much Improved: number analyzed (Participants) | 39 | 4 | 11 | 29
  Week 12: Much Improved | 28.2 | 75.0 | 36.4 | 41.4
  Week 12: Very Much Improved: number analyzed (Participants) | 39 | 4 | 11 | 29
  Week 12: Very Much Improved | 5.1 | 25.0 | 0 | 10.3
  Week 18: Improved: number analyzed (Participants) | 36 | 4 | 11 | 29
  Week 18: Improved | 36.1 | 25.0 | 27.3 | 31.0
  Week 18: Much Improved: number analyzed (Participants) | 36 | 4 | 11 | 29
  Week 18: Much Improved | 25.0 | 50.0 | 54.5 | 41.4
  Week 18: Very Much Improved: number analyzed (Participants) | 36 | 4 | 11 | 29
  Week 18: Very Much Improved | 11.1 | 25.0 | 9.1 | 13.8

7. Secondary Outcome: Change From Baseline in 36-item Short-Form Health Survey (SF-36)
Description: Change from baseline to Week 12 in SF-36 is reported. The SF-36 assesses 8 health concepts: 1) limitations in physical activities because of health problems (physical functioning); 2) limitations in social activities because of physical or emotional problems (social functioning); 3) limitations in usual role activities because of physical health problems (role physical); 4) bodily pain; 5) general mental health; 6) limitations in usual role activities because of emotional problems (role emotional); 7) vitality; and 8) general health perceptions. The items use Likert-type scales with either 5 or 6 points, or 2 or 3 points. Higher SF-36 scores indicate a better state of health. The score for a section is an average of the individual question scores, which are scaled 0-100 (100=highest level of functioning).
Time Frame: Baseline (Day -7 to Day -1, inclusive) and Week 12
Population: mITT population included all participants who received at least 1 dose of any double-blind study drug and have at least 1 daily NRS assessment while receiving the treatment. Number of participants analyzed (N) denotes the number of participants evaluated for this outcome measure.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | MEDl7352 Low Dose | MEDl7352 Meduim Dose | MEDI7352 High Dose
Number analyzed (Participants) | 39 | 4 | 12 | 29
Units on a scale
  Physical Functioning | 11.282 (17.0412) | 21.248 (13.1526) | 0.417 (19.7084) | 12.759 (16.6141)
  Role Physical | 7.372 (18.0159) | 28.125 (27.7169) | 0.000 (37.3101) | 6.681 (17.4338)
  Bodily Pain | 8.3 (20.51) | 9.8 (22.75) | 12.1 (23.11) | 14.9 (17.30)
  General Health | -2.6 (17.70) | -2.5 (5.00) | -5.3 (17.72) | 0.0 (19.98)
  Vitality | -0.160 (20.6039) | 3.125 (16.5359) | -0.521 (17.7695) | -4.095 (24.0486)
  Social Functioning | 1.92 (19.772) | 31.25 (23.936) | -1.04 (24.108) | 9.05 (23.121)
  Role Emotional | -1.923 (25.3248) | 8.333 (31.9110) | -5.556 (34.8748) | -1.724 (19.9681)
  Mental Health | -5.9 (21.82) | 10.0 (20.41) | -1.3 (14.48) | -0.7 (18.41)

8. Secondary Outcome: Percentage of Participants Taking Any Rescue Medication
Description: Percentage of participants taking any rescue medication are reported. Participants were asked to record all rescue medications they take for neuropathic pain in a paper diary.
Time Frame: Baseline (Day -7 to Day -1, inclusive) through Week 12
Population: mITT population included all participants who received at least 1 dose of any double-blind study drug and have at least 1 daily NRS assessment while receiving the treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | MEDl7352 Low Dose | MEDl7352 Meduim Dose | MEDI7352 High Dose
Number analyzed (Participants) | 54 | 4 | 14 | 35
Percentage of participants | 13 | 0 | 14.3 | 8.6

9. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Treatment Emergent Serious Adverse Events (TESAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. The TEAEs are defined as events present at baseline that worsened in intensity after administration of study drug or events absent at baseline that emerged after administration of study drug.
Time Frame: Day 1 through 20.42 weeks (maximum observed duration)
Population: Safety population included all participants who received at least 1 dose of any double-blind study drug and were analyzed according to the treatment they actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MEDl7352 Low Dose | MEDl7352 Meduim Dose | MEDI7352 High Dose
Number analyzed (Participants) | 54 | 4 | 14 | 35
Participants
  Any TEAEs | 30 | 4 | 10 | 23
  Any TESAEs | 1 | 0 | 0 | 0

10. Secondary Outcome: Number of Participants With Abnormal Vital Signs Reported as TEAEs
Description: Number of participants with abnormal vital signs reported as TEAEs are reported. Abnormal vital signs are defined as any abnormal finding in the vital sign parameters (body temperature, diastolic blood pressure, systolic blood pressure, heart [pulse] rate, and respiratory rate).
Time Frame: Day 1 through 20.42 weeks (maximum observed duration)
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MEDl7352 Low Dose | MEDl7352 Meduim Dose | MEDI7352 High Dose
Number analyzed (Participants) | 54 | 4 | 14 | 35
Participants
  Blood pressure increased | 0 | 0 | 0 | 1
  Hypotension | 0 | 0 | 0 | 1
  Hypertension | 1 | 0 | 0 | 0
  Orthostatic hypertension | 1 | 0 | 0 | 0
  Orthostatic hypotension | 3 | 0 | 0 | 0

11. Secondary Outcome: Number of Participants With Clinically Significant Abnormal Electrocardiograms (ECGs)
Description: Number of participants with clinically significant abnormal ECGs are reported.
Time Frame: Day 1 through 20.42 weeks (maximum observed duration)
Population: Safety population included all participants who received at least 1 dose of any double-blind study drug and were analyzed according to the treatment they actually received. Number of participants analyzed (N) denotes the number of participants who were evaluable for the specified outcome measure. Here, number analyzed (n) denotes those participants who were evaluable at the specified time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MEDl7352 Low Dose | MEDl7352 Meduim Dose | MEDI7352 High Dose
Number analyzed (Participants) | 54 | 4 | 14 | 35
Participants
  Day 1 | 1 | 0 | 0 | 0
  Week 4: number analyzed (Participants) | 50 | 4 | 13 | 32
  Week 4 | 0 | 0 | 1 | 0
  Week 8: number analyzed (Participants) | 45 | 4 | 12 | 32
  Week 8 | 0 | 0 | 0 | 1
  Week 12: number analyzed (Participants) | 40 | 4 | 11 | 31
  Week 12 | 1 | 0 | 0 | 1
  Week 18 (follow-up): number analyzed (Participants) | 40 | 4 | 12 | 30
  Week 18 (follow-up) | 0 | 0 | 1 | 0

12. Secondary Outcome: Number of Participants With Abnormal Clinical Laboratory Parameters Reported as TEAEs
Description: Number of participants with abnormal clinical laboratory parameters reported as TEAEs are reported. Abnormal clinical laboratory parameters defined as any abnormal finding during analysis of hematology, clinical chemistry, coagulation, and urinalysis.
Time Frame: Day 1 through 20.42 weeks (maximum observed duration)
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MEDl7352 Low Dose | MEDl7352 Meduim Dose | MEDI7352 High Dose
Number analyzed (Participants) | 54 | 4 | 14 | 35
Participants
  Alanine aminotransferase increased | 0 | 0 | 2 | 0
  Blood glucose decreased | 0 | 0 | 1 | 1
  Aspartate aminotransferase increased | 0 | 0 | 1 | 0
  Blood glucose increased | 0 | 0 | 0 | 1
  C-reactive protein increased | 1 | 0 | 0 | 1
  Coagulation test abnormal | 0 | 0 | 0 | 1
  Glomerular filtration rate decreased | 0 | 0 | 0 | 1
  White blood cells urine positive | 0 | 0 | 0 | 1
  Bacterial test positive | 1 | 0 | 0 | 0
  Blood bilirubin increased | 1 | 0 | 0 | 0
  Protein urine present | 1 | 0 | 0 | 0
  Urine analysis abnormal | 1 | 0 | 0 | 0
  Hypoglycemia | 1 | 0 | 1 | 1
  Hypercholesterolaemia | 0 | 0 | 0 | 1
  Hyperglycaemia | 1 | 0 | 1 | 0

13. Secondary Outcome: Number of Participants With Clinically Significant Findings in Physical Examination Reported as TEAEs
Description: Number of participants with clinically significant findings in physical examination reported as TEAE are reported. A complete physical examination (excluding the genitourinary examination, unless warranted) was performed.
Time Frame: Day 1 through 20.42 weeks (maximum observed duration)
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MEDl7352 Low Dose | MEDl7352 Meduim Dose | MEDI7352 High Dose
Number analyzed (Participants) | 54 | 4 | 14 | 35
Participants | 1 | 0 | 0 | 1

14. Secondary Outcome: Number of Participants With Clinically Significant Findings in Neurological Examination
Description: Number of participants with clinically significant findings in neurological examination is reported.
Time Frame: Day 1 through 20.42 weeks (maximum observed duration)
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MEDl7352 Low Dose | MEDl7352 Meduim Dose | MEDI7352 High Dose
Number analyzed (Participants) | 54 | 4 | 14 | 35
Participants | 0 | 0 | 0 | 0

15. Secondary Outcome: Number of Participants With Abnormal Dorsiflexion Strength
Description: Number of participants with abnormal dorsiflexion strength is reported. Dorsiflexion strength is scored on 0-4 scale. The scale indicated 0 = normal power, 1 = mild weakness, 2 = moderate weakness, 3 = severe weakness, and 4 = paralysis.
Time Frame: Day 1 through 20.42 weeks (maximum observed duration)
Population: Safety population included all participants who received at least 1 dose of any double-blind study drug and were analyzed according to the treatment they actually received. Here, number of participants analyzed (N) denotes those participants who were assessed for strength and deep tendon reflexes assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MEDl7352 Low Dose | MEDl7352 Meduim Dose | MEDI7352 High Dose
Number analyzed (Participants) | 40 | 4 | 12 | 30
Participants
  Mild Weakness | 9 | 0 | 7 | 18
  Moderate Weakness | 8 | 0 | 0 | 2
  Severe Weakness | 0 | 0 | 0 | 0
  Paralysis | 0 | 0 | 0 | 0

16. Secondary Outcome: Number of Participants With Abnormal Deep Tendon Reflex (Knee and Ankle)
Description: Number of participants with abnormal deep tendon reflex are reported. Deep tendon reflex (knee and ankle) strength is scored on 0-4 scale. The scale indicated 0 = normal, 1 = ankle reflex reduced, 2 = ankle reflex absent, 3 = ankle reflex absent and knee reflex reduced, and 4 = all reflexes (both ankle and knee) absent. Participants within a specific row are not included in any other row in the data table below.
Time Frame: Day 1 through 20.42 weeks (maximum observed duration)
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MEDl7352 Low Dose | MEDl7352 Meduim Dose | MEDI7352 High Dose
Number analyzed (Participants) | 40 | 4 | 12 | 30
Participants
  Ankle reflex reduced | 5 | 2 | 2 | 3
  Ankle reflex absent | 4 | 0 | 1 | 5
  Ankle reflex absent and knee reflex reduced | 11 | 1 | 3 | 13
  All reflexes absent | 15 | 0 | 6 | 5

17. Secondary Outcome: Change From Baseline in Total Neuropathy Score-Nurse (TNSn)
Description: The TNSn, a semi-quantitative clinical assessment of peripheral nervous system function, was administered at baseline (Screening), Day 1, Weeks 2, 4, 6, 8, 10, 12 and Week 18/early termination. The TNSn provides for an assessment of motor symptom score, autonomic symptom score, pin sensibility score, and vibration sensibility score. Each neuropathy item is scored on a 0-4 scale. The scores are summed to obtain a total score ranging from 0 to 20. Higher total scores correlate with more severe neuropathy. Not all of the early terminated participants completed the 18 week assessment. Only 3 early terminated participants contributed data at the Week 18 assessment.
Time Frame: Baseline (Day -45 to -1), pre-dose on Day 1, Weeks 2, 4, 6, 8, 10, 12, and 18/early termination
Population: Safety population included all participants who received at least 1 dose of any double-blind study drug and were analyzed according to the treatment they actually received. Number of participants analyzed (N) denotes the number of participants evaluated for this outcome measure. Here, number analyzed (n) denotes those participants who were evaluable at the specified time point.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | MEDl7352 Low Dose | MEDl7352 Meduim Dose | MEDI7352 High Dose
Number analyzed (Participants) | 50 | 4 | 13 | 34
Units on a scale
  Day 1: number analyzed (Participants) | 4 | 0 | 0 | 1
  Day 1 | -0.25 (0.957) |  |  | 1.00 (NA) — Standard deviation was not reported as only one participant was evaluable for this arm
  Week 2: number analyzed (Participants) | 48 | 4 | 13 | 34
  Week 2 | -0.54 (1.304) | -1.25 (1.258) | 0.00 (1.354) | -0.94 (2.117)
  Week 4: number analyzed (Participants) | 50 | 4 | 13 | 32
  Week 4 | -0.90 (1.982) | -2.50 (3.786) | -0.85 (1.819) | -1.19 (1.891)
  Week 6: number analyzed (Participants) | 45 | 4 | 12 | 33
  Week 6 | -1.40 (2.071) | -0.75 (2.872) | -1.00 (1.859) | -1.85 (2.093)
  Week 8: number analyzed (Participants) | 45 | 4 | 12 | 32
  Week 8 | -1.40 (2.082) | -2.50 (3.000) | -0.92 (1.881) | -1.84 (2.665)
  Week 10: number analyzed (Participants) | 40 | 4 | 12 | 31
  Week 10 | -1.90 (2.458) | -2.00 (3.916) | -1.67 (1.435) | -2.45 (3.042)
  Week 12: number analyzed (Participants) | 40 | 4 | 12 | 30
  Week 12 | -1.73 (2.562) | -2.25 (2.062) | -2.17 (1.899) | -2.53 (2.515)
  Week 18: number analyzed (Participants) | 40 | 4 | 12 | 30
  Week 18 | -2.00 (2.631) | -2.50 (3.512) | -2.17 (2.329) | -2.30 (3.053)

18. Secondary Outcome: Number of Participants With Investigator Reported Significant Changes From Baseline in Motor and Sensory Nerve Conduction
Description: Motor and sensory nerve conduction studies were performed in relevant lower and upper limb nerves (sural, peroneal, median/ulnar, fibular, and tibial nerves) wherein amplitude, peak latency, conduction velocity, and duration of nerve action potentials were recorded.
Time Frame: Day 1 through 20.42 weeks (maximum observed duration)
Population: Safety population included all participants who received at least 1 dose of any study drug and were analyzed according to the treatment they actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MEDl7352 Low Dose | MEDl7352 Meduim Dose | MEDI7352 High Dose
Number analyzed (Participants) | 54 | 4 | 14 | 35
Participants | 2 | 0 | 0 | 0

19. Secondary Outcome: Number of Participants With at Least One Concomitant Medication
Description: Number of participants with at least one concomitant medication is reported. A concomitant medication is defined as any medication continuing or starting after first dose of study medication.
Time Frame: Day 1 through 20.42 weeks (maximum observed duration)
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MEDl7352 Low Dose | MEDl7352 Meduim Dose | MEDI7352 High Dose
Number analyzed (Participants) | 54 | 4 | 14 | 35
Participants | 54 | 4 | 14 | 35

20. Secondary Outcome: Number of Participants With Injection Site Reaction
Description: Number of participants with injection site reaction is reported.
Time Frame: Day 1 through 20.42 weeks (maximum observed duration)
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MEDl7352 Low Dose | MEDl7352 Meduim Dose | MEDI7352 High Dose
Number analyzed (Participants) | 54 | 4 | 14 | 35
Participants | 1 | 1 | 0 | 0

21. Secondary Outcome: Number of Participants With Infusion Reaction
Description: Number of participants with infusion reaction is reported.
Time Frame: Day 1 through 20.42 weeks (maximum observed duration)
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MEDl7352 Low Dose | MEDl7352 Meduim Dose | MEDI7352 High Dose
Number analyzed (Participants) | 54 | 4 | 14 | 35
Participants | 0 | 0 | 0 | 2

22. Secondary Outcome: Serum Total Nerve Growth Factor (NGF) Concentrations
Description: Serum concentrations of total NGF in ADA positive or negative participants are reported.
Time Frame: Day 1 (pre-dose; baseline), Weeks 2, 4, 6, 8, 10 (Day 70; pre-dose, immediately before end of infusion, 8 hours and 24 hours post Day 70 infusion [Day 71]), 11, and 12 (approximately same time of day as Week 10 infusion)
Population: Safety population: participants received at least 1 dose of any double-blind study drug and were analyzed according to treatment actually received. Number of participants analyzed: participants evaluated for this outcome measure. Number analyzed (n): participants evaluable at specified time point. MEDl7352 low and medium dose group data is not reported due to change in assay during course of study and stability data not supporting re-analysis of early study samples with new in-house assay.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Placebo | MEDl7352 Low Dose | MEDl7352 Meduim Dose | MEDI7352 High Dose
Number analyzed (Participants) | 30 | 0 | 0 | 31
pg/mL
  Day 1 | 52.303 (11.6178) |  |  | 65.687 (60.4036)
  Week 2: number analyzed (Participants) | 29 | 0 | 0 | 29
  Week 2 | 62.613 (15.1088) |  |  | 2384.760 (1989.0309)
  Week 4: number analyzed (Participants) | 29 | 0 | 0 | 29
  Week 4 | 78.209 (92.0122) |  |  | 2213.699 (2408.3112)
  Week 6: number analyzed (Participants) | 27 | 0 | 0 | 29
  Week 6 | 64.661 (18.6478) |  |  | 2361.855 (2645.8141)
  Week 8: number analyzed (Participants) | 26 | 0 | 0 | 29
  Week 8 | 63.291 (16.5332) |  |  | 1992.129 (2507.9826)
  Week 10 (pre-dose): number analyzed (Participants) | 25 | 0 | 0 | 28
  Week 10 (pre-dose) | 173.383 (563.8921) |  |  | 1681.073 (2455.0666)
  Week 10 (before end of infusion): number analyzed (Participants) | 25 | 0 | 0 | 28
  Week 10 (before end of infusion) | 57.308 (13.3588) |  |  | 1992.756 (2968.1285)
  Week 10 (8 hours post-dose): number analyzed (Participants) | 25 | 0 | 0 | 28
  Week 10 (8 hours post-dose) | 177.323 (554.8131) |  |  | 2012.384 (2795.8138)
  Week 10 (post 24 hours): number analyzed (Participants) | 24 | 0 | 0 | 28
  Week 10 (post 24 hours) | 222.980 (772.9408) |  |  | 1849.835 (2671.9526)
  Week 11: number analyzed (Participants) | 25 | 0 | 0 | 26
  Week 11 | 59.441 (13.6892) |  |  | 1743.100 (2621.0687)
  Week 12: number analyzed (Participants) | 25 | 0 | 0 | 28
  Week 12 | 63.416 (18.4243) |  |  | 1710.966 (2838.0975)

23. Secondary Outcome: Number of Participants With Positive Anti-Drug Antibodies (ADA) to MEDI7352
Description: Number of participants with positive ADA to MEDI7352 are reported. Treatment-induced ADA positive is defined as ADA negative at baseline and positive at least 1 post-baseline assessment. Treatment-boosted ADA positive is defined as ADA positive at baseline with pre-existing titre boosted by 4-fold or greater during the study period. Persistent positive is defined as ADA negative at baseline and positive at least 2 post-baseline assessments (with >= 16 weeks between first and last positive) or ADA positive at last post-baseline assessment. Transiently positive is defined as ADA negative at baseline and at least one post-baseline ADA positive measurement and not fulfilling the conditions for persistently positive.
Time Frame: Pre-dose at baseline (Day -45 to -1) and Study Weeks 2, 4, 8, 10, 12, and 18 (follow-up)
Population: Safety population included all participants who received at least 1 dose of any double-blind study drug and were analyzed according to the treatment they actually received. Here, number of participants analyzed (N) denotes those participants who had adequate ADA sample.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MEDl7352 Low Dose | MEDl7352 Meduim Dose | MEDI7352 High Dose
Number analyzed (Participants) | 53 | 4 | 14 | 35
Participants
  Treatment-induced ADA | 0 | 3 | 7 | 28
  Treatment-boosted ADA | 0 | 0 | 1 | 1
  Persistently positive ADA | 0 | 3 | 6 | 26
  Transiently positive ADA | 0 | 0 | 1 | 2

ADVERSE EVENTS:
Time Frame: Day 1 through 20.42 weeks (maximum observed duration)
Description: Safety population included all participants who received at least 1 dose of any double-blind study drug and were analyzed according to the treatment they actually received.
Arm/Group | Placebo | MEDl7352 Low Dose | MEDl7352 Meduim Dose | MEDI7352 High Dose
All-Cause Mortality (participants affected / at risk) | 0/54 | 0/4 | 0/14 | 0/35
Serious Adverse Events (participants affected / at risk) | 1/54 | 0/4 | 0/14 | 0/35
Other Adverse Events (participants affected / at risk) | 30/54 | 4/4 | 10/14 | 23/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=54) | MEDl7352 Low Dose (N=4) | MEDl7352 Meduim Dose (N=14) | MEDI7352 High Dose (N=35)
Lung abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=54) | MEDl7352 Low Dose (N=4) | MEDl7352 Meduim Dose (N=14) | MEDI7352 High Dose (N=35)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 4 (5)
Urinary tract infection (Infections and infestations) | 2 (3) | 0 (0) | 2 (2) | 1 (1)
Nasopharyngitis (Infections and infestations) | 11 (11) | 0 (0) | 0 (0) | 2 (3)
Acute sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 5 (9) | 3 (24) | 1 (2) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (4) | 0 (0) | 1 (1)
Allodynia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Burning sensation (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Orthostatic intolerance (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetic neuropathy (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Sensory disturbance (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Blood glucose decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
C-reactive protein increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Coagulation test abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Glomerular filtration rate decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
White blood cells urine positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bacterial test positive (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymph node palpable (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Protein urine present (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urine analysis abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 5 (6) | 0 (0) | 0 (0) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Frequent bowel movements (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Change of bowel habit (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia oral (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (3)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
Soft tissue mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (3) | 0 (0) | 1 (1) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hand dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lichenification (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Skin burning sensation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Catheter site swelling (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Facial pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site reaction (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Feeling hot (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gravitational oedema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Nail injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Repetitive strain injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrioventricular block first degree (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Conjunctival hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye irritation (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retinal haemorrhage (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphoedema (Vascular disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Orthostatic hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bruxism (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract inflammation (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Dose-response relationship outcome was not evaluated by MCP-MOD because of insufficient number of doses. The study was prematurely terminated due to longer enrolment time than was anticipated. A combined population PK analysis was reported separately from the main CSR as a stand-alone report.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AstraZeneca has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.

DOCUMENTS (2):
  • Study Protocol (2022-04-13): https://cdn.clinicaltrials.gov/large-docs/34/NCT03755934/Prot_002.pdf
  • Statistical Analysis Plan (2023-10-04): https://cdn.clinicaltrials.gov/large-docs/34/NCT03755934/SAP_003.pdf